CLINICAL TRIAL: NCT02891382
Title: Feasibility Study on the Impact of Economic Incentives for Weight Loss to Improve the Management of Type 2 Diabetes Mellitus: REDEEM Feasibility Study
Brief Title: Feasibility Study on the Impact of Economic Incentives to Improve the Management of Type 2 Diabetes Mellitus
Acronym: REDEEM-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MR/M007405/1
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Weight Loss; Financial Incentives; Hemoglobin A, Glycosylated
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Weight Loss | interventions — Organizational Objectives

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Individual incentives - Arm 1 (Experimental): This arm receives diabetes education + goal setting + individual rewards
  Interventions: Behavioral: Diabetes education; Behavioral: Goal setting; Behavioral: Individual Reward
- Mixed incentives (Altruism) - Arm 2 (Experimental): This arm receives diabetes education + goal setting + companion support + individual rewards
  Interventions: Behavioral: Diabetes education; Behavioral: Goal setting; Behavioral: Companion Support; Behavioral: Individual Reward
- Mixed Incentives (Cooperation) - Arm 3 (Experimental): This arm receives diabetes education + goal setting + companion support + shared rewards
  Interventions: Behavioral: Diabetes education; Behavioral: Goal setting; Behavioral: Companion Support; Behavioral: Shared Reward

INTERVENTIONS:
Behavioral: Diabetes education — Participants interact with a diabetes educator (DE), every two weeks.
Behavioral: Goal setting — Goals for weight loss and change in levels of HbA1c
Behavioral: Companion Support — Patient has a companion/team support partner to support achieving goals.
  Arms: Mixed Incentives (Cooperation) - Arm 3; Mixed incentives (Altruism) - Arm 2
Behavioral: Individual Reward — The cash reward is given to the patient with diabetes.
  Arms: Individual incentives - Arm 1; Mixed incentives (Altruism) - Arm 2
Behavioral: Shared Reward — Patients with diabetes and their companion support will each receive 50% of the cash reward.
  Arms: Mixed Incentives (Cooperation) - Arm 3

SUMMARY:
This feasibility study aims to compare the implementation process of three different interventions that use economic incentives to promote lifestyle behavioral changes in patients with type 2 diabetes mellitus, and to identify barriers and facilitators linked to the process of implementing each of the interventions. The interventions are based on economic incentives directed to the patient (individual incentives) or a team comprised by the patient and a partner (mixed incentives).

Design: Three-month randomized control feasibility study to test the feasibility of implementing three types of intervention with economic incentives in patients with diabetes mellitus.

Setting: Diabetes outpatient clinics from a public hospital in Peru.

DETAILED DESCRIPTION:
Economic incentives have been used to promote changes in habits such as smoking and weight loss. However, no studies have been done to determine the impact of this strategy on the management of type 2 diabetes mellitus (T2DM). Additionally, previous studies do not describe ways to determine the amount of an economic incentive to promote behavioral changes, e.g adherence to treatment, increased physical activity and adherence to a healthy diet. There are also questions regarding the frequency of incentives, the type of incentive (cash or other prizes), and the preferred payment method that this study will allow us to explore. Furthermore, we want to test whether a "team work approach" (mixed incentives) vs. an "individual approach" (individual incentives) can also play a role in introducing behavioral changes.

The goal of the study is to learn about the implementation process of three different interventions that use economic incentives to promote behavioral changes in patients with T2DM, and identify main barriers and facilitators tied to the implementation process of each intervention.

This feasibility study will provide key insights to inform a future larger study; specifically, we will

* Learn about the experience of participants with T2DM with economic incentives.
* Learn about the experience of the companion/team support partners of the participants with T2DM.
* Evaluate the patient's receptiveness to and comprehension of the educational materials used to promote behavioral changes.
* Evaluate the patient and the companion/team support partner's receptiveness towards the received economic incentive as a tool for promoting behavioral changes.
* Explore the companion/team support partner's activities that are most effective in helping with T2DM management of patients.
* Explore whether patients with T2DM are able to keep a daily record of their efforts to manage their diabetes.
* Evaluate the feasibility of packaging and implementing a future clinical trial that evaluates the impact of the use of economic incentives and teamwork in people with T2DM.

From a clinical perspective, we will evaluate the feasibility of reaching the proposed clinical goals in terms of weight loss and HbA1c levels after the intervention period.

Interventions

Diabetes education (all arms). In the introductory meeting, a diabetes educator will explain to the participants all the procedures, including details of the number of sessions, and the participant's received a manual with information about diabetes management with a tailored weight loss plan. Each participant will be offered up to seven follow- up sessions with the diabetes educator, every two weeks, plus a final session, thus totaling up to 9 one-to-one interactions during the trial, provided that the participant attended all of their meetings. Participants will also be provided with a logbook to register their efforts regarding introducing changes in diet and physical activity. The information from this logbook will provide the starting point for conversations with the diabetes educator during the follow-up sessions, every two weeks.

Goal setting (all arms). To determine eligibility for a cash reward, three goals were pre-specified: (1) Weight loss, 80 PEN if the participant loses one kilogram over a period of two weeks, (2) HbA1c level, 200 PEN if the participant achieves, at the end of the study, a decrease in 1% compared to their baseline level, and (3) HbA1c level and control, 400 PEN if the participant achieves, at the end of the study, a decrease ≥1% of A1c or reaches levels of A1c ≤6.5% compared to their baseline level. At the end of the study, targets for weight loss and HbA1c were evaluated independently, i.e. participants could receive more than one reward provided that each independent target was achieved.

Companion/team support (Arm 2 and Arm 3). A companion/team support for each participant also receives information about diabetes care in the initial session and a brochure to guide and support the treatment process of the participant. The activities of the companion/team support member will be recorded, and they will be offered to join the follow- up sessions with the patient, every two weeks, but these will not be compulsory.

Cash rewards. Two types of rewards will be considered. (1) Individual rewards (Arm 1 and Arm 2), the reward will be provided to the participant. If the participant were to have a companion/team support partner, the cash reward was given to the participant and no rules about sharing the reward (or not) with their companion/team support are established. (2) Shared rewards (Arm 3), i.e. the participant and their companion/team support will receive 50% of the cash reward each.

ELIGIBILITY:
Inclusion criteria for participants:

* Type 2 diabetes mellitus
* Body mass index 25-39.9 kg/m2, irrespective of HbA1c status
* Able to give consent

Exclusion Criteria for participants:

* Diagnosis of cancer or another serious comorbidity
* Pharmacotherapy for weight loss or corticosteroids
* Pregnant women
* Blindness, amputation, foot ulcer or being on dialysis
* Be companion/team support for another participant in the trial

Inclusion criteria for the companion/team support:

* Available and committed to supporting the participant in achieving their goals
* Able to provide consent

Exclusion criteria for the companion/team support:

* Physical or mental condition that does not allow him to help the participant to achieve goals

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-07; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Miranda, MD, PhD, Principal Investigator — Universidad Peruana Cayetano Heredia; Antonio Trujillo, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Hospital Nacional Arzobispo Loayza, Lima, Peru

IPD SHARING:
Plan to Share IPD: Yes
Following on MRC's data sharing policy, we plan to make our quantitative datasets available in platforms for data sharing (e.g. Figshare, etc.). Qualitative data will be available upon request.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: The dataset with quantitative information will be available within six months from the publication of the main manuscript.
Access Criteria: Contact cronicas@oficinas-upch.pe; maria.pesantes.v@upch.pe; maria.lazo@upch.pe; and/or jaime.miranda@upch.pe
URL: https://www.mrc.ac.uk/research/policies-and-guidance-for-researchers/data-sharing/

REFERENCES:
- [Result] Pesantes MA, Del Valle A, Diez-Canseco F, Bernabe-Ortiz A, Portocarrero J, Trujillo A, Cornejo P, Manrique K, Miranda JJ. Family Support and Diabetes: Patient's Experiences From a Public Hospital in Peru. Qual Health Res. 2018 Oct;28(12):1871-1882. doi: 10.1177/1049732318784906. Epub 2018 Aug 1. PMID 30066604
- [Derived] Miranda JJ, Lazo-Porras M, Bernabe-Ortiz A, Pesantes MA, Diez-Canseco F, Cornejo SDP, Trujillo AJ. The effect of individual and mixed rewards on diabetes management: A feasibility randomized controlled trial. Wellcome Open Res. 2019 Feb 5;3:139. doi: 10.12688/wellcomeopenres.14824.3. eCollection 2018. PMID 30662958
- See also: REVISED A descriptive study of potential participant preferences for the design of an incentivised weight loss programme for people with type 2 diabetes mellitus attending a public hospital in Lima, Peru — https://wellcomeopenresearch.org/articles/3-53/v2
- See also: The effect of individual and mixed rewards on diabetes management: A feasibility randomized controlled trial — https://wellcomeopenresearch.org/articles/3-139/v1
- Available data/document: Individual Participant Data Set — https://figshare.com/articles/REDEEM_Study_Feasibility_pilot_study/7180802

RESULTS

PARTICIPANT FLOW:
Groups:
- Mixed Incentives (Altruism) - Arm 2 Patients: This arm receives diabetes education + goal setting + companion support + individual rewards
  Diabetes education: Participants interact with a diabetes educator (DE), every two weeks.
  Goal setting: Goals for weight loss and change in levels of HbA1c
  Companion Support: Patient has a companion/team support partner to help him/her in achieving goals.
  Individual Reward: The cash reward is given to the patient with diabetes.
- Mixed Incentives (Altruism) - Arm 2 Companions: The companion support help the partner to achieve goals.
  The cash reward is given to the patient with diabetes and not to the companion.
- Mixed Incentives (Cooperation) - Arm 3 Patients: This arm receives diabetes education + goal setting + companion support + shared rewards
  Diabetes education: Participants interact with a diabetes educator (DE), every two weeks.
  Goal setting: Goals for weight loss and change in levels of HbA1c
  Companion Support: Patient has a companion/team support partner to help him/her in achieving goals.
  Shared Reward: Patients with diabetes and their companion support will each receive 50% of the cash reward.
- Mixed Incentives (Cooperation) - Arm 3 Companions: The companion support help the partner to achieve goals.
  Patients with diabetes and their companion support will each receive 50% of the cash reward.
Period: Overall Study
Arm/Group | Individual Incentives - Arm 1 | Mixed Incentives (Altruism) - Arm 2 Patients | Mixed Incentives (Altruism) - Arm 2 Companions | Mixed Incentives (Cooperation) - Arm 3 Patients | Mixed Incentives (Cooperation) - Arm 3 Companions
Started | 18 | 18 (These participants have their companions) | 18 | 18 (These participants have their companions) | 18
Completed | 15 | 14 | 13 | 15 | 14
Not Completed | 3 | 4 | 5 | 3 | 4
Not completed — Lost to Follow-up | 3 | 4 | 5 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Mixed Incentives (Altruism) - Arm 2 Patients: This arm receives diabetes education + goal setting + companion support + individual rewards
  Diabetes education: Participants interact with a diabetes educator (DE), every two weeks.
  Goal setting: Goals for weight loss and change in levels of HbA1c
  Companion Support: Patient has a companion/team support partner to support achieving goals.
  Individual Reward: The cash reward is given to the patient with diabetes.
- Mixed Incentives (Cooperation) - Arm 3 Patient: This arm receives diabetes education + goal setting + companion support + shared rewards
  Diabetes education: Participants interact with a diabetes educator (DE), every two weeks.
  Goal setting: Goals for weight loss and change in levels of HbA1c
  Companion Support: Patient has a companion/team support partner to support achieving goals.
  Shared Reward: Patients with diabetes and their companion support will each receive 50% of the cash reward.
- Mixed Incentives (Cooperation) - Arm 3 Companion: The companion support help the partner to achieve goals.
  Patients with diabetes and their companion support will each receive 50% of the cash reward.
- Total: Total of all reporting groups
Arm/Group | Individual Incentives - Arm 1 | Mixed Incentives (Altruism) - Arm 2 Patients | Mixed Incentives (Altruism) - Arm 2 Companions | Mixed Incentives (Cooperation) - Arm 3 Patient | Mixed Incentives (Cooperation) - Arm 3 Companion | Total
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 15 | 16 | 18 | 81
  >=65 years | 2 | 2 | 3 | 2 | 0 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (9.8) | 55.5 (9.8) | 49.8 (15.9) | 54.2 (7.6) | 39.7 (16.6) | 54.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 11 | 12 | 11 | 58
  Male | 6 | 6 | 7 | 6 | 7 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 18 | 18 | 18 | 18 | 18 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Peru | 18 | 18 | 18 | 18 | 18 | 90
Glycated Hemoglobin [Mean (Standard Deviation); unit: "Percentage of glycated hemoglobin"] — Percentage of glycated hemoglobin at baseline Population: Glycated hemoglobin was not analyzed in the companions
  "Percentage of glycated hemoglobin"
    number analyzed (Participants) | 18 | 18 | 0 | 18 | 0 | 54
    (all) | 8.5 (2.2) | 7.9 (3.1) |  | 8.2 (2.1) |  | 8.2 (2.5)
Weight [Mean (Standard Deviation); unit: Kg] — Weight at baseline Population: Clinical data was not measure in the companions
  Kg
    number analyzed (Participants) | 18 | 18 | 0 | 18 | 0 | 54
    (all) | 76.9 (10.7) | 84.5 (17.4) |  | 85.1 (22.3) |  | 82.1 (17.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Hemoglobin
Description: HbA1c change at 3 months from baseline
Time Frame: Baseline and 3 months
Population: Some participants had data about weight but not about glycated hemoglobin and for that reason the number of participants in this table are different from the table that show the results of weight.
Measure: Mean (Standard Deviation); unit: "Percentage of glycated hemoglobin"
Arm/Group | Individual Incentives - Arm 1 | Mixed Incentives (Altruism) - Arm 2 | Mixed Incentives (Cooperation) - Arm 3
Number analyzed (Participants) | 13 | 13 | 14
"Percentage of glycated hemoglobin" | 1.4 (1.4) | 0.9 (1.2) | 1.1 (1.6)

2. Secondary Outcome: Change in Weight
Description: Weight change at 3 months from baseline
Time Frame: Baseline and 3 months
Population: Some participants had data about weight but not about glycated hemoglobin and for that reason the number of participants in this table are different from the table that show the results of glycated hemoglobin.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Individual Incentives - Arm 1 | Mixed Incentives (Altruism) - Arm 2 | Mixed Incentives (Cooperation) - Arm 3
Number analyzed (Participants) | 15 | 14 | 15
Kg | 2.9 (2.2) | 0.4 (2.5) | 0.4 (3.0)

ADVERSE EVENTS:
Time Frame: 3 months
Description: The intervention implemented in the participants had low risk of serious adverse events. For that reason we applied a non-systematic assessment.
  Also, adverse events were not monitored/assessed for the companions.
Groups:
- Mixed Incentives (Cooperation) - Arm 3 Patients: This arm receives diabetes education + goal setting + companion support + shared rewards
  Diabetes education: Participants interact with a diabetes educator (DE), every two weeks.
  Goal setting: Goals for weight loss and change in levels of HbA1c
  Companion Support: Patient has a companion/team support partner to support achieving goals.
  Shared Reward: Patients with diabetes and their companion support will each receive 50% of the cash reward.
Arm/Group | Individual Incentives - Arm 1 | Mixed Incentives (Altruism) - Arm 2 Patients | Mixed Incentives (Cooperation) - Arm 3 Patients
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT02891382/Prot_SAP_000.pdf